CLINICAL TRIAL: NCT07175857
Title: Evaluation of the Efficacy of an Innovative Digital Therapeutic Medical Device, Lyv Endo, for the Management of Patients With Endometriosis
Acronym: LYVENDO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lyv Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LYVENDO
Record Dates: First submitted 2025-08-07; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Endometriosis
Keywords: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): standard care
- Intervention (Experimental): Use of the Lyv Endo app + standard care
  Interventions: Device: Lyv Endo app

INTERVENTIONS:
Device: Lyv Endo app — Lyv Endo is a CE-marked Class I therapeutic digital medical device offering a patient-centered, integrative approach. Its innovation lies in its ability to deliver personalized content based on symptoms, surpassing the limits of traditional care.
  Arms: Intervention

SUMMARY:
The main objective of this clinical study is to evaluate the clinical impact of using an innovative digital therapeutic device on the quality of life of patients with endometriosis.

The working hypothesis is that the therapeutic digital medical device Lyv Endo may improve quality of life and reduce symptom intensity by enhancing patient engagement in the management of their condition. This justifies the need to evaluate the effect of Lyv Endo as a complement to standard medical care.

DETAILED DESCRIPTION:
Endometriosis is a chronic, systemic, and inflammatory disease. Long considered a gynecological condition, endometriosis is now recognized as a systemic disease associated with symptoms and comorbidities that extend well beyond the reproductive system, affecting psychological well-being, social life, and professional activity. Endometriosis affects nearly 10% of women of reproductive age, corresponding to an estimated 1.5 to 2.5 million women in France. It is most commonly diagnosed in women aged 25 to 49 years, who represent 68.3% of cases, whereas women under 25 are rarely diagnosed (fewer than 4%). According to the French Haute Autorité de Santé (HAS), the prevalence of endometriosis may affect between 600,000 and 700,000 women aged 18 to 50 years in France.

Endometriosis is characterized by the presence of endometrium-like tissue outside the uterus, which may lead to severe pain, particularly during menstruation, as well as infertility in approximately one-third of cases. On average, diagnosis is delayed by seven years, complicating the management of the disease. Common symptoms include severe menstrual pain (dysmenorrhea), chronic pelvic pain, deep dyspareunia, dyschezia during menstruation, cyclic urinary symptoms, and infertility.

Diagnosis is primarily clinical, supported by imaging examinations such as transvaginal ultrasound and pelvic MRI to confirm the presence of lesions. In the absence of conclusive findings, empirical treatment may be initiated based on symptom relief, with a presumptive diagnosis. Laparoscopy, previously a routine diagnostic procedure, is now reserved for complex cases where imaging is inconclusive and treatments have failed.

To date, there is no curative treatment for endometriosis. Current treatments are symptomatic and include hormonal therapies (progestins or combined oral contraceptives), hormonal intrauterine devices, and analgesics (e.g., tramadol, nefopam, paracetamol-codeine or paracetamol-tramadol combinations). Up to 83% of patients continue to experience persistent symptoms despite medical or surgical treatment. In cases of severe pain or infertility resistant to treatment, surgical intervention may be considered, although recurrence is possible.

Given the chronic nature of the symptoms, endometriosis is a complex, multifactorial disease requiring multidisciplinary care. An integrative approach-including therapeutic education, regular physical activity, psychological support, and dietary measures-is essential to improve symptom management and patient quality of life. Supportive therapies such as physiotherapy and sophrology have shown benefits in endometriosis patients. These non-pharmacological therapies are increasingly recommended by pain specialists to address central sensitization and help raise pain thresholds, which are pathologically low in patients with chronic pelvic pain. This multimodal and multidisciplinary approach, as a complement to conventional pharmacological treatment, aligns with the HAS recommendations for managing chronic pain, which apply to endometriosis patients.

However, most patients still lack access to such multidisciplinary care. This gap may be partly due to insufficient training in endometriosis among frontline healthcare professionals (e.g., general practitioners and community gynecologists), who are often unaware of the proven benefits of this type of approach and do not refer patients to relevant professionals (e.g., physiotherapists, psychologists, sex therapists). Additionally, the number of healthcare professionals specialized in endometriosis remains limited, especially in medically underserved areas. Finally, due to limited consultation time, healthcare providers may not be able to address all these aspects during routine visits.

Over the past decade, the development of digital technologies and connected devices has opened new perspectives in patient care. These tools can play a crucial role by offering innovative solutions to relieve pain, enhance patient education, and foster greater autonomy in symptom self-management. In the field of endometriosis, there are currently very few digital medical devices specifically dedicated to supporting patients.

The Lyv Endo device is a CE-marked Class I digital therapeutic medical device that stands out through its integrative, patient-centered approach to endometriosis management. Its innovation lies in its ability to deliver comprehensive and personalized content tailored to each patient's symptoms, addressing key limitations of traditional care (e.g., limited consultation time, low availability of trained professionals). This digital medical device offers individualized therapeutic support across five key modules: disease knowledge, mental well-being, adapted physical activity, nutrition, and sexual health. Lyv Endo is positioned at the forefront of digital medical technologies, with the goal of transforming endometriosis care.

The main objective is to evaluate the clinical impact of using an innovative digital therapeutic device on the quality of life of patients with endometriosis.

Secondary Objectives :

* To evaluate the clinical impact of using the Lyv Endo digital therapeutic on the quality of life of patients with endometriosis
* To evaluate the clinical impact on symptoms and complications associated with endometriosis
* To evaluate the clinical impact on mental health
* To assess the impact on lifestyle habits
* To assess the organizational impact
* To assess the health economic impact
* To evaluate the usability of the full version of the therapeutic digital medical device

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years old
* with confirmed endometriosis diagnosis
* symptomatic patients (NRS ≥ 4 on one or more symptoms)
* French-speaking
* Owning a smartphone with internet/data,
* covered by French social security

Exclusion Criteria:

* Planned surgery during the study or surgery in the past 8 weeks
* Fertility hormone treatment during study
* Previous use of full Lyv Endo app or pilot program
* Pregnant or breastfeeding
* Under legal protection (guardianship, etc.)
* Cognitive or psychiatric conditions compromising consent
* Judged non-autonomous by investigator
* Participation in another interventional study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 304 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Clinical impact | Baseline and 3 months
  Change in Endometriosis Health Profile-5 score ranging from 0 (best outcome) to 100 (worst outcome)

SECONDARY OUTCOMES:
Clinical Impact | Baseline and 3 months
  Change in Quality of Life : variation in EuroQol 5-Dimension (EQ-5D-5L) ranging from level 1(no problem) to level 5 (unable to/extreme problems)
Clinical Impact | 3 months
  Change in Quality of Life: proportion of patients with deterioration of quality of life based on Endometriosis Health Profile-5 (EHP-5) total score (MCID = 4.5 points)
Clinical Impact | Baseline and 3 months
  Change in global symptom intensity: variation in total and subgroup Numeric Rating Scale scores (0 = best outcome; 10 = worst outcome)
Clinical Impact | Baseline and 3 months
  Change in Sensitization: variation in Central sensitization inventory (CSI) ranging from 0 (best outcome) to 36 (worst outcome)
Clinical Impact | Baseline and 3 months
  Change in depression level: variation in Patient Health Questionnaire-9 (PHQ-9) scores (0 = best outcome; 27 = worst outcome)
Clinical Impact | Baseline and 3 months
  Change in anxiety level: variation in Generalized Anxiety Disorder-7 (GAD-7) scores (0 = best outcome; 21 = worst outcome)
Clinical Impact | From baseline to 3 months
  Change in associated analgesic consumption: monthly evolution of analgesic use
Clinical Impact | Baseline and 3 months
  Change in lifestyle habits: frequency of physical activity
Clinical Impact | Baseline and 3 months
  Change in lifestyle habits: percentage of patients with adapted eating behaviors
Clinical Impact | Baseline and 3 months
  Change in lifestyle habits: sleep quality
Organisational Impact | Baseline and 3 months
  Change in organisational parameters: number of endometriosis-related healthcare visits
Organisational Impact | Baseline and 3 months
  Change in organisational parameters: duration of sick leaves
Organisational Impact | Baseline and 3 months
  Change in organisational parameters: variation in Work Productivity and Activity Impairment questionnaire (WPAI) scores (0 = best outcome; 10 = worst outcome)
Health Economic impact | 3 months
  Comparative analysis of health economic parameters: cost-utility analysis
Health Economic impact | 3 months
  Description: Comparative analysis of health economic parameters: estimated costs for the French National Health Insurance
Health Economic Impact | 3 months
  Comparative analysis of health economic parameters: healthcare resource utilization
Usability of Therapeutic Digital Medical Device | From Baseline to 3 months
  Adherence rate
Usability of Therapeutic Digital Medical Device | From Baseline to 3 months
  Number of logins
Usability of Therapeutic Digital Medical Device | From Baseline to 3 months
  Engagement with the personalized program
Usability of Therapeutic Digital Medical Device | 3 months
  Satisfaction level and System Usability Scale (SUS) score (0 = worst outcome; 100 = best outcome)

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Clinique Tivoli Ducos, Bordeaux
  - Centre Hospitalier de Versailles, Le Chesnay
  - Centre Hospitalier Le Mans, Le Mans
  - Hôpital Le Blois, Lille
  - Hôpital Paris Saint-Joseph, Paris
  - Centre Hospitalier de Saint Nazaire, Saint-Nazaire

REFERENCES:
- [Background] Breton Z, Stern E, Pinault M, Lhuillery D, Petit E, Panel P, Alexaline M. A Digital Program for Daily Life Management With Endometriosis: Pilot Cohort Study on Symptoms and Quality of Life Among Participants. JMIR Form Res. 2025 Feb 28;9:e58262. doi: 10.2196/58262. PMID 39791286
- [Background] Aubry G, Panel P, Thiollier G, Huchon C, Fauconnier A. Measuring health-related quality of life in women with endometriosis: comparing the clinimetric properties of the Endometriosis Health Profile-5 (EHP-5) and the EuroQol-5D (EQ-5D). Hum Reprod. 2017 Jun 1;32(6):1258-1269. doi: 10.1093/humrep/dex057. PMID 28383700
- [Background] O'Hara R, Rowe H, Fisher J. Managing endometriosis: a cross-sectional survey of women in Australia. J Psychosom Obstet Gynaecol. 2022 Sep;43(3):265-272. doi: 10.1080/0167482X.2020.1825374. Epub 2020 Oct 13. PMID 33050751
- [Background] Coxon L, Vollert J, Perro D, Lunde CE, Ferreira-Gomes J, Charrua A, Abreu-Mendes P, Krassowski M, Birch J, Meijlink J, Hummelshoj L, Hoffmann A, Aziz Q, Arendt-Nielsen L, Pogatzki-Zahn E, Evans E, Demetriou L, McMahon SB, Missmer SA, Becker CM, Zondervan KT, Horne AW, Cruz F, Sieberg CB, Treede RD, Nagel J, Vincent K. Comprehensive quantitative sensory testing shows altered sensory function in women with chronic pelvic pain: results from the Translational Research in Pelvic Pain (TRiPP) Study. Pain. 2023 Nov 1;164(11):2528-2539. doi: 10.1097/j.pain.0000000000002955. Epub 2023 Jun 7. PMID 37289573
- [Background] Cohen SP, Vase L, Hooten WM. Chronic pain: an update on burden, best practices, and new advances. Lancet. 2021 May 29;397(10289):2082-2097. doi: 10.1016/S0140-6736(21)00393-7. PMID 34062143
- [Background] Zondervan KT, Becker CM, Missmer SA. Endometriosis. N Engl J Med. 2020 Mar 26;382(13):1244-1256. doi: 10.1056/NEJMra1810764. No abstract available. PMID 32212520
- See also: Description of the Lyv Endo app in french — https://www.lyv.app/application